CLINICAL TRIAL: NCT00959855
Title: Long-term Evaluation of Activity and Health Status Pre and Post Pulmonary Rehabilitation - A Multi-Centred Trial.
Brief Title: Long-term Impact of Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Collaborators: ITS Pulmonary Rehabilitation Research Network (Unknown)
Responsible Party: Principal Investigator, Professor Richard Costello, consultant chest physician, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ITS-1-MCT
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary Rehabilitation; Inflammation; Oxidative Stress; Steps; Free Living Activities; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary Rehabilitation (Experimental): Pulmonary rehabilitation classes based on the British Thoracic Society guidelines will be undertaken for two hours for 16 sessions within an eight week period.
  Interventions: Other: Pulmonary Rehabilitation
- Pulmonary Rehabiliation (No Intervention): The control group will be assessed in the same time frame without participating in the rehabilitation class. They will avail of the next available class after the 12 month assessment.

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Sixteen, two hourly pulmonary rehabilitation sessions over an eight week period. The first hour will consist of an individualized exercise programme based on exercise field tests. The second hour will consist of an educational component. A home exercise programme of inspiratory muscle training (Threshold(R)IMT (respiratory muscle trainer re:HS730EU-001 single patient use) starting between 15% -30% of PiMax and progress weekly to 60% for 30 mins a day/ 5 dats a week with an inspiratory/expiratory ratio of 3:4. Patients will also be encouraged to walk or undertake an home exercise programme based on a Borg score of between 3 and 5 an additional 3 days a week.
  Other Names: Activity Armbands; Inspiratory Muscle Training
  Arms: Pulmonary Rehabilitation

SUMMARY:
This study has been designed to capture a large group of patients who undergo pulmonary rehabilitation and map their progression over a 5 year time-frame.

The outcome measures have been chosen to capture physiological, functional capacity, free-living activities plus admission and exacerbation rates thereby enhancing our understanding of the potential effects exercise and self management techniques may have on the disease progression.

Pulmonary rehabilitation has not been shown to reduce inflammation; therefore, unlike acute exacerbation's where a decrease in inflammation indicates recovery, the exact mechanisms responsible for improvement during pulmonary rehabilitation are as yet unknown.

DETAILED DESCRIPTION:
The benefits of pulmonary rehabilitation are well documented elsewhere, however, the exact mechanisms responsible for these significant improvements and alteration of the disease progression are unexplained. Also unexplained is the apparent lack of carry over of functional capacity into free-living activities as measured by activity monitors.

There are no reported effects on decreasing level of inflammatory cytokines or C-reactive protein (CRP) post rehabilitation, however, a training response to reactive oxidative stress (ROS) after a moderate intensity pulmonary rehabilitation programme has been reported. As oxidative stress is a catalyst to inflammation, a training response to exercise induced ROS in patients with COPD may also have a secondary effect of modifying inflammation in the stable COPD patient thereby improving patient outcomes.

No studies to-date have combined free-living activities, biomarkers and standard outcome measures in patient's pre and post pulmonary rehabilitation or follow-up patients over a five year period.

Subjects referred to pulmonary rehabilitation who fulfil the GOLD criteria for COPD will be recruited on a rolling basis and randomly allocated to one of two groups. Group 1 (Control), Group 2 (Intervention).

It is a multi-centred, randomised controlled trial using the above convenience sample of patients referred to pulmonary rehabilitation who meet the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of COPD based on the GOLD staging of the Disease
2. MMRC score of 3 or above
3. Ability to mobilize independently
4. Willing to comply with the home exercise and inspiratory muscle training programmes
5. Willing to wear the SenseWare Armband
6. Optimal medical management
7. No adverse effects to exercise testing
8. Patient's awaiting lung transplant

Exclusion Criteria:

1. Evidence of ischemic heart disease/acute changes on ECG
2. Uncontrolled hypertension
3. Insulin dependent diabetes mellitus
4. Uncontrolled CCF / idiopathic cardiomyopathy
5. Reversible Asthma
6. A diagnosis of lung cancer/TB/recent pneumothorax/PE or pneumonia
7. Any musculoskeletal/neurological condition which would render the patient incapable of completing the course
8. Exacerbation of COPD within 4 weeks of program
9. Poor cognitive status
10. Previous attendance at a pulmonary rehabilitation program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Quality of life score | One year
  St George's quality of life score at the end of one year will be compared between those who underwent rehabilitaion and those who were in the control non intervention group.

SECONDARY OUTCOMES:
Spiromtery | 12 months
  Differences between the intervention group at 12 months .
Number of exacerbations of COPD. | over one year
  The number of exacerbations of COPD will be compared between the control and the rehabilitation group.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Costello, Professor, Principal Investigator — Beaumont Hosptial
Locations (1):
- Beaumont Hospital, Beaumont, Dublin, Ireland